CLINICAL TRIAL: NCT05541185
Title: Effects of Nigella Sativa Oil on Pain Intensity and Physical Functions in Patients With Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Effects of Nigella Sativa Oil on Pain Intensity and Physical Functions in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan ÇEÇEN (Other)
Responsible Party: Sponsor-Investigator, Sultan ÇEÇEN, Lecturer, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Nigella Sativa Oil
Record Dates: First submitted 2022-08-28; First posted 2022-09-15 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
Keywords: Nursing; Osteoarthritis; Nigella sativa; Pain; Massage
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Nigella sativa oil; Naproxen; Massage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nigella sativa oil group (Experimental): 1 ml of nigella sativa oil was applied to both knee areas of the nigella sativa oil group by massaging for 2 minutes three times a day for 21 days.
  Interventions: Biological: Nigella sativa oil
- Naproxen and lidocaine gel group (Experimental): 1 ml of naproxen and lidocaine gel was applied to both knee areas of the naproxen and lidocaine gel group by massaging for 2 minutes three times a day for 21 days.
  Interventions: Biological: Naproxen and lidocaine gel
- Massage group (Placebo Comparator): 1 ml of vaseline was applied to both knee areas of the massage group by massaging for 2 minutes three times a day for 21 days.
  Interventions: Biological: Massage

INTERVENTIONS:
Biological: Nigella sativa oil — 1 ml of nigella sativa oil was applied to both knee areas of the nigella sativa oil group by massaging for 2 minutes three times a day for 21 days.
  Arms: Nigella sativa oil group
Biological: Naproxen and lidocaine gel — 1 ml of Naproxen and lidocaine gel was applied to both knee areas of the Naproxen and lidocaine gel group by massaging for 2 minutes three times a day for 21 days.
  Arms: Naproxen and lidocaine gel group
Biological: Massage — 1 ml of vaseline was applied to both knee areas of the massage group by massaging for 2 minutes three times a day for 21 days.
  Arms: Massage group

SUMMARY:
Purpose: The study was conducted to determine the effect of 1 ml of nigella sativa oil applied for 2 minutes three times a day for 21 days on pain severity and physical functions in patients with knee osteoarthritis (OA).

Design and methods: This randomized controlled study was conducted with patients diagnosed with knee OA and admitted to the physical therapy outpatient clinic of a public hospital in Turkey between February 15, 2021 and March 31, 2021. A total of 75 patients were included in the study, and 25 of them were assigned to the nigella sativa oil group, 25 to the naproxen and lidocaine gel group, and 25 to the massage group. Research data were collected using the "Patient Information Form", "Western Ontario and McMaster Universities Osteoarthritis Index (Western Ontario and McMaster Universities Osteoarthritis Index = WOMAC)" and knee joint range measurements were made. For 21 days, both knees were massaged for 2 minutes 3 times a day, 1 ml of nigella sativa oil was applied to the patients in the nigella sativa oil group, 1 ml of naproxen and lidocaine gel was applied to the patients in the naproxen and lidocaine gel group, and 1 ml of liquid vaseline was applied to the patients in the massage group.

DETAILED DESCRIPTION:
Osteoarthritis (OA); It is a chronic degenerative joint disease that is frequently seen in all societies due to many factors such as age, gender, genetics, osteoporosis, high activity level, diet, obesity and occupation, negatively affecting the quality of life and causing problems such as joint pain and limitation of movement in the affected joint. Articular cartilage, subchondral bone, synovial membrane and periarticular muscles as well as all joint structures are affected by this disease. According to the Health Research data conducted by the Turkish Statistical Institute in 2019, it was determined that 14.6% of women over the age of 15, 7.6% of men and 11.2% of the general total had arthritis problems in Turkey. The World Health Organization estimates that 18% of women over the age of 60 and 9.6% of men worldwide experience OA symptoms, 80% of them develop limitation of movement due to pain and loss of function, and 25% are unable to perform activities of daily living. OA, whose incidence and prevalence increases with aging in particular, affects the knee, waist, neck, hip and hand at a high rate, while it affects the shoulder and ankle at a low rate. Common complaints; joint pain, stiffness, edema on the joint, a feeling of being stuck with the movement of the joint, and decreased range of motion. It is stated that the condition that most affects the patient is pain and psychological changes related to the disease.

Since current medical treatment approaches cannot prevent tissue degeneration in OA, relief of pain and improvement of joint functions are at the forefront of treatment. In this respect, integrative approaches consisting of pharmacological, non-pharmacological and surgical or a combination of these are used in the treatment.

In pharmacological treatment, starting with paracetamol according to the severity of the pain and increasing the severity of pain, non-steroidal anti-inflammatory drugs (NSAIDs), COX-2 inhibitors, and topical drugs are switched. In addition, in some selected cases, intra-articular steroid and hyaluronic acid injections and centrally acting analgesic drugs are also preferred. However, it is stated that these drugs should be used with caution in terms of their efficacy and side effects, and gastrointestinal and renal side effects are more common in long-term use of NSAIDs, especially in elderly individuals.

Rest, regular aerobics, muscle strengthening and range of motion exercises, aquatic exercise, transcutaneous electrical nerve stimulation, crutches, walker, cane, corset, elastic bandage, insoles and appropriate shoes use, weight loss as well as joint protection of the patient and coping with the disease. Education about methods constitutes non-pharmacological treatment. In surgical treatment, osteotomy, arthroscopy and, as a last resort, arthroplasty are performed in patients with persistent pain whose activities of daily living are severely restricted. In the Consensus Report of the Turkish Rheumatism Research and Combat Association (2012), evidence-based recommendations for the treatment of knee OA; It is stated that integrative treatments can be used in addition to pharmacological and non-pharmacological treatments, provided that they are monitored in terms of their effects and side effects. In the literature, it has been observed that integrative treatments such as massage therapy, herbal treatments, balneotherapy, acupuncture, and Tai chi are effective for OA.

It is stated that among the integrated treatments, especially herbal medicines have been used in articular diseases for 2000 years and they do not have any side effects, and in recent years, medicinal plants have become a new source of medicine due to many side effects of synthetic drugs. One of these medicinal herbal remedies is nigella sativa oil, which belongs to the Ranunculaceae family, commonly known as black cumin in traditional medicine. The active nutraceutical ingredient of the oil is thymoquinone. Nigella sativa oil is rich in unsaturated fatty acids such as oleic acid and can relieve pain by inhibiting the activity of the cyclooxygenase enzyme, as well as showing anti-inflammatory, antidiabetic, anticonvulsant, anticancer, anti-aging, immunomodulator, antimicrobial, spasmolytic, bronchodilator, hepatoprotective, renoprotective, gastroprotective and antioxidant effects. is also indicated.

A limited number of studies have been found in the literature indicating that nigella sativa oil reduces pain and improves physical function in patients with OA. Therefore, in this study, it was aimed to examine the effect of 1 ml of nigella sativa oil applied with massage for 2 minutes three times a day for 21 days on pain severity and physical functions in patients with knee OA and to contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* - 50 years or older,
* Can speak Turkish and have no communication problems,
* Diagnosed with knee OA by the physician according to the ACR criteria, and grade 2-3 according to the radiological classification of Kellgren and Lawrence,
* Having knee pain in the last three months and needing analgesics more than 15 days in a month,
* Does not use gel for analgesic purposes locally on the knee area,
* Able to walk
* Having crepitus in motion,
* No inflammatory disease
* No history of malignancy,
* Does not have an open wound in the application area,
* No known allergic condition to Nigella sativa oil, naproxen and lidocaine gel and vaseline,
* Patients without any psychiatric disorders were included in the study

Exclusion Criteria:

* - under the age of 50,
* Blindness or deafness
* Does not speak Turkish and cannot be communicated,
* Any disease that cannot be cured,
* Having a physical disability in the area where the application will be made,
* Any skin disease in the area to be treated,
* Having large scar tissue in the area to be treated,
* Having a history of physical trauma in the last three months in the area to be treated,
* Any peripheral vascular disease in the area to be treated,
* With inflammatory joint disease,
* Having a history of rheumatoid arthritis and fibromyalgia,
* Using any complementary and integrative (integrated) health application in the last three months,
* Those who have been treated with drugs into the joint in the last three months,
* Receiving pain blocking therapy in the last year,
* Receiving physical therapy in the last three months and during the application,
* Using antipsychotic, narcotic and corticosteroids,
* Patients with different analgesic use or irregular drug use were not included in the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
1st Measurement | first day
  In the first measurement, "Western Ontario and McMaster Universities Osteoarthritis Index" were applied to the patients included in the Nigella sativa oil, naproxen and lidocaine gel and massage groups. The scores that can be obtained from the scale are 0-20 for pain, 0-8 for stiffness, and 0-68 for difficulty in performing daily physical activities. Higher scores indicate more symptoms and increased physical limitation.

SECONDARY OUTCOMES:
2nd Measurement/ seventh day | seventh day
  The second measurement was obtained by reapplying Western Ontario and McMaster Universities Osteoarthritis Index .
  The scores that can be obtained from the scale are 0-20 for pain, 0-8 for stiffness, and 0-68 for difficulty in performing daily physical activities. Higher scores indicate more symptoms and increased physical limitation.

OTHER OUTCOMES:
3rd Measurement | the fourteenth day
  The third measurement was obtained by reapplication of Western Ontario and McMaster Universities Osteoarthritis Index.
  The scores that can be obtained from the scale are 0-20 for pain, 0-8 for stiffness, and 0-68 for difficulty in performing daily physical activities. Higher scores indicate more symptoms and increased physical limitation.
4th Measurement | twenty-first day
  Western Ontario and McMaster Universities Osteoarthritis Index was applied for the last time and the 4th measurement results were obtained by evaluating the knee joint range with a goniometer.
  The scores that can be obtained from the scale are 0-20 for pain, 0-8 for stiffness, and 0-68 for difficulty in performing daily physical activities. Higher scores indicate more symptoms and increased physical limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participation data will be made available for all outcome measures.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Kooshki A, Forouzan R, Rakhshani MH, Mohammadi M. Effect of Topical Application of Nigella Sativa Oil and Oral Acetaminophen on Pain in Elderly with Knee Osteoarthritis: A Crossover Clinical Trial. Electron Physician. 2016 Nov 25;8(11):3193-3197. doi: 10.19082/3193. eCollection 2016 Nov. PMID 28344755
- [Background] Huseini HF, Kianbakht S, Mirshamsi MH, Zarch AB. Effectiveness of Topical Nigella sativa Seed Oil in the Treatment of Cyclic Mastalgia: A Randomized, Triple-Blind, Active, and Placebo-Controlled Clinical Trial. Planta Med. 2016 Mar;82(4):285-8. doi: 10.1055/s-0035-1558208. Epub 2015 Nov 19. PMID 26584456